CLINICAL TRIAL: NCT02261467
Title: Evaluation of the Safety and Efficacy of Treatment With BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for Subjects With Forehead and Glabellar Facial Rhytides
Brief Title: A Safety and Efficacy Study of OnabotulinumtoxinA in Forehead and Glabellar Facial Rhytides
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-142; 2014-001860-36 (EudraCT Number)
Record Dates: First submitted 2014-10-03; First posted 2014-10-10 (Estimated); Results first posted 2017-06-23 (Actual); Last update posted 2019-01-08 (Actual); Status verified 2018-12

CONDITIONS: Forehead Rhytides; Glabellar Rhytides
MeSH Terms: interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OnabotulinumtoxinA (Experimental): OnabotulinumtoxinA injected into the protocol-specified areas on Day 1. Subjects will receive at least 1 and up to 3 treatments.
  Interventions: Biological: OnabotulinumtoxinA
- Placebo followed by OnabotulinumtoxinA in Period 2 (Placebo Comparator): Placebo (normal saline) injected into the protocol-specified areas on Day 1. If the subject meets the re-treatment criteria in Period 2, the subject will receive up to 2 open-label treatments with onabotulinumtoxinA into the protocol-specified areas.
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Biological: OnabotulinumtoxinA — OnabotulinumtoxinA injected into the protocol-specified areas. Subjects will receive at least 1 and up to 3 treatments.
  Other Names: BOTOX® Cosmetic; botulinum toxin Type A
  Arms: OnabotulinumtoxinA
Drug: Normal Saline — Placebo (normal saline) injected into the protocol-specified areas on Day 1.
  Arms: Placebo followed by OnabotulinumtoxinA in Period 2

SUMMARY:
This is a safety and efficacy study of onabotulinumtoxinA in subjects with forehead and glabellar facial rhytides (frown lines).

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe forehead and glabellar lines
* Willing to have facial photos taken

Exclusion Criteria:

* Prior exposure to botulinum toxin of any serotype for any indication
* Anticipated need for treatment with botulinum toxin of any serotype for any indication during the study, other than study treatment
* Diagnosis of myasthenia gravis, Eaton-Lambert syndrome, or amyotrophic lateral sclerosis
* Any facial resurfacing laser or light treatment, microdermabrasion, or superficial peels in the past 3 months
* Any medium depth or deep depth facial chemical peels; facial skin resurfacing; or permanent facial make-up in the past 6 months
* Any nonpermanent soft tissue fillers, or treatment with oral retinoids in the past year
* Prior face lift, thread lift, eyebrow lift, or related procedures (eg, eyelid and/or eyebrow surgery)
* Prior facial treatment with permanent soft tissue fillers, synthetic implants (eg, Gore-Tex®), and/or fat transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2014-10-21 (Actual); Primary Completion 2015-06-04 (Actual); Study Completion 2016-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (16):
- United States (9):
  - Total Skin and Beauty Dermatology Center, PC, Birmingham, Alabama
  - Advanced Research Associates, Glendale, Arizona
  - Clinical Science Institute, Santa Monica, California
  - About Skin Dermatology and DermSurgery, PC, Greenwood Village, Colorado
  - Steven Fagien, MD, PA, Boca Raton, Florida
  - Laser & Skin Surgery Center of Indiana, Carmel, Indiana
  - Coleman Center For Cosmetic Dermatologic Surgery, Metairie, Louisiana
  - Henry Ford Medical Center, West Bloomfield, Michigan
  - NW Dermatology and Research Center, Portland, Oregon
- Canada (5):
  - Carruthers Dermatology Centre, Vancouver, British Columbia
  - Dr. Shannon Humphrey, Inc., Vancouver, British Columbia
  - Jean Carruthers Cosmetic Dermatology, Vancouver, British Columbia
  - Sweat Clinics of Canada, Toronto, Ontario
  - Arthur Swift Research, Inc., Westmount, Quebec
- Ireland (2):
  - Aesthetic Surgery Ireland, Dublin
  - Beacon Face and Dermatology Clinic, Dublin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] De Boulle K, Werschler WP, Gold MH, Bruce S, Sattler G, Ogilvie P, Street J, Larsen KE, Yushmanova I, Lei X, Lee E, Vitarella D, Mao C. Phase 3 Study of OnabotulinumtoxinA Distributed Between Frontalis, Glabellar Complex, and Lateral Canthal Areas for Treatment of Upper Facial Lines. Dermatol Surg. 2018 Nov;44(11):1437-1448. doi: 10.1097/DSS.0000000000001612. PMID 30096106

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 421 subjects were enrolled in the study, of these, 30 subjects were excluded from the data analyses at one site. The participant flow reflects all subjects included in the data analyses.
Pre-assignment Details: Subjects were randomized to either placebo or onabotulinumtoxinA in Period 1. Subjects randomized to receive placebo in Period 1 who subsequently received open-label onabotulinumtoxinA in Period 2 are also included in the onabotulinumtoxinA group for the Safety analysis.
Period: Overall Study
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Started | 101 | 290
Completed | 80 | 253
Not Completed | 21 | 37
Not completed — Enrolled in Error | 1 | 0
Not completed — Protocol Violation | 0 | 1
Not completed — Personal Reasons | 17 | 22
Not completed — Lost to Follow-up | 2 | 13
Not completed — Adverse Event | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA | Total
Number analyzed (Participants) | 101 | 290 | 391
Age, Customized [Number; unit: Participants]
  <65 years | 101 | 281 | 382
  >=65 years | 0 | 9 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 87 | 249 | 336
  Male | 14 | 41 | 55

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With ≥2-Grade Improvement From Baseline on Both the Investigator's and Subject's Facial Wrinkle Scale (FWS) Ratings of Forehead Line Severity at Maximum Eyebrow Elevation
Description: The Investigator and subject each assessed the severity of the subject's forehead lines at maximum eyebrow elevation using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with at least a 2-grade improvement from baseline assessed by both the Investigator and the subject are reported.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 101 | 290
Percentage of Subjects | 0.0 [NA to NA] — Zero incidences; therefore, CI not applicable | 61.4 [55.8 to 67.0]

2. Secondary Outcome: Percentage of Subjects With an Investigator Rating of None or Mild on the 4-Grade FWS for Forehead Line Severity at Maximum Eyebrow Elevation
Description: The Investigator assessed the severity of the subject's forehead lines at maximum eyebrow elevation using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with a score of "none" and "mild" are reported.
Time Frame: Day 30
Population: Intent-to-Treat: all randomized subjects with a score of "none" and "mild" on the FWS at maximum eyebrow elevation
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 101 | 290
Percentage of Subjects | 2.0 [-0.7 to 4.7] | 94.1 [91.4 to 96.8]

3. Secondary Outcome: Percentage of Subjects With ≥1-Grade Improvement From Baseline on the Investigator's FWS Rating of Forehead Line Severity at Rest
Description: The Investigator assessed the severity of the subject's forehead lines at rest using the 4-grade FWS, where 0=none, 1=mild, 2=moderate, and 3=severe. The percentage of subjects with at least a 1-grade improvement assessed by the Investigator are reported.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with at least a 1-grade improvement assessed by the Investigator on the FWS at rest
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 96 | 278
Percentage of Subjects | 19.8 [11.8 to 27.8] | 85.6 [81.5 to 89.7]

4. Secondary Outcome: Percentage of Subjects Reporting Mostly Satisfied or Very Satisfied on the 5-Point Facial Line Satisfaction Questionnaire (FLSQ) Item 5
Description: The FLSQ consists of 13 questions that assess subject satisfaction and appearance-related impacts associated with facial lines. Item 5 on the FLSQ asks "How satisfied are you with the effect your treatment had on your facial lines?" Responses included: very satisfied, mostly satisfied, neither satisfied or dissatisfied, mostly dissatisfied, or very dissatisfied. The percentage of subjects reporting a score of mostly satisfied or very satisfied with treatment are reported.
Time Frame: Day 60
Population: Intent-to-Treat: all randomized subjects with data reported at this time point
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 99 | 289
Percentage of Subjects | 1.0 [-1.0 to 3.0] | 90.3 [86.9 to 93.7]

5. Secondary Outcome: Percentage of Subjects With ≥20-Point Improvement From Baseline on the Impact Domain of the FLSQ Among Subjects With Baseline Score ≥ 20 Points
Description: The FLSQ consists of 13 questions that assess subject satisfaction and appearance-related impacts associated with facial lines. The Impact Domain measures the subject's appearance-related and emotional impacts of treatment and is composed of 5 questions with a possible range of scores from 0 (worst) to 100 (best), using a transformed scale. Only subjects with baseline scores ≥ 20 are included in the analysis.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with baseline scores ≥ 20 on the Impact Domain of the FLSQ
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 90 | 268
Percentage of Subjects | 18.9 [10.8 to 27.0] | 73.9 [68.6 to 79.1]

6. Secondary Outcome: Percentage of Subjects With a ≥3-Point Improvement From Baseline on Item 4 of the 11-Point Facial Line Outcomes (FLO-11) Questionnaire©
Description: The FLO-11 assess the subject's psychological and appearance-related impacts associated with facial lines. Item 4 is "I look older than my actual age because of my facial lines" with a range of possible scores from 0 = not at all to 10 = very much. Only subjects with baseline scores ≥ 3 are included in the analysis.
Time Frame: Baseline, Day 30
Population: Intent-to-Treat: all randomized subjects with baseline scores ≥ 3 on Item 4 of the FLO-11
Measure: Number (95% Confidence Interval); unit: Percentage of Subjects
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 89 | 246
Percentage of Subjects | 11.2 [4.7 to 17.8] | 77.2 [72.0 to 82.5]

7. Secondary Outcome: Time to Retreatment Eligibility
Description: Time to retreatment eligibility is defined as the number of days from treatment cycle 1 injection to the return to an Investigator FWS rating of moderate or severe at maximum eyebrow elevation. The FWS is a 4-grade scale, where 0=none, 1=mild, 2=moderate, and 3=severe. Only subjects who achieved a ≥ 2-grade improvement on both the Investigator and subject FWS ratings at maximum eyebrow elevation on Day 30 are included in the analysis.
Time Frame: 12 Months
Population: Intent-to-Treat: all randomized subjects who achieved a ≥ 2-grade improvement on both the Investigator and subject FWS ratings at maximum eyebrow elevation
Measure: Median (Standard Deviation); unit: Days
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Number analyzed (Participants) | 0 | 174
Days |  | 119 (52.9)

ADVERSE EVENTS:
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess adverse events and serious adverse events. Subjects randomized to receive placebo in Period 1 who subsequently received open-label onabotulinumtoxinA in Period 2 are included in the onabotulinumtoxinA group for the Safety analysis.
Arm/Group | Placebo Followed by OnabotulinumtoxinA in Period 2 | OnabotulinumtoxinA
Serious Adverse Events (participants affected / at risk) | 0/100 | 5/374
Other Adverse Events (participants affected / at risk) | 12/100 | 92/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Followed by OnabotulinumtoxinA in Period 2 (N=100) | OnabotulinumtoxinA (N=374)
Angina pectoris (Cardiac disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Followed by OnabotulinumtoxinA in Period 2 (N=100) | OnabotulinumtoxinA (N=374)
Injection site bruising (General disorders) | 2 | 19
Nasopharyngitis (Infections and infestations) | 3 | 30
Headache (Nervous system disorders) | 7 | 43

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.